CLINICAL TRIAL: NCT00334750
Title: Distribution of Risk Factors Amongst Ocular Hypertension and Open-Angle Glaucoma Patients in Canada
Brief Title: Distribution of Risk Factors in Ocular Hypertension and Open-Angle Glaucoma Patients in Canada
Status: Completed | Type: Observational
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Other Study IDs: A6111125
Record Dates: First submitted 2006-06-05; First posted 2006-06-08 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2010-09

CONDITIONS: Glaucoma, Open-Angle; Ocular Hypertension
Keywords: Glaucoma, Open-Angle Ocular Hypertension Risk factors Canadian
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- There is no intervention in this study: This study is collecting information on the presence of risk factors in new diagnosed OH and OAG patients in Canada.
  Interventions: Other: There is no intervention in this study.

INTERVENTIONS:
Other: There is no intervention in this study. — This study is collecting information on the presence of risk factors in new diagnosed OH and OAG patients in Canada.

SUMMARY:
This descriptive, non-interventional study will collect information on the presence of risk factors in newly diagnosed ocular hypertension and open-angle glaucoma patients in Canada.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed at study visit or within 3 months of visit with OH
* OAG (to include POAG, NTG, pigmentary and pseudoexfoliation glaucoma)

Exclusion Criteria:

* No prior treatment for OH or OAG
* No prior ocular surgery or history of ocular trauma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Canadian population
Sampling Method: Non-Probability Sample
Enrollment: 410 (Actual)
Dates: Start 2007-11; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
To describe the presence and distribution of risk factors in subjects diagnosed with OH or OAG stratified according to geographic distribution in a Canadian population in the ophthalmologist practice. | duration of study

SECONDARY OUTCOMES:
To describe the severity of disease at the time of diagnosis and to determine if there is a correlation between risk factors, or number of risk factors, and the severity of disease at presentation. | duration of study

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (16):
- Canada (16):
  - Pfizer Investigational Site, Calgary, Alberta
  - Pfizer Investigational Site, Edmonton, Alberta
  - Pfizer Investigational Site, Nanaimo, British Columbia
  - Pfizer Investigational Site, Vancouver, British Columbia
  - Pfizer Investigational Site, Williams Lake, British Columbia
  - Pfizer Investigational Site, Winnipeg, Manitoba
  - Pfizer Investigational Site, Sydney, Nova Scotia
  - Pfizer Investigational Site, Brampton, Ontario
  - Pfizer Investigational Site, Hamilton, Ontario
  - Pfizer Investigational Site, London, Ontario
  - Pfizer Investigational Site, Mississauga, Ontario
  - Pfizer Investigational Site, Oakville, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Montreal, Quebec
  - Pfizer Investigational Site, Sherbrooke, Quebec
  - Pfizer Investigational Site, Saskatoon, Saskatchewan

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6111125&StudyName=Distribution%20of%20risk%20factors%20in%20Ocular%20Hypertension%20and%20Open-Angle%20Glaucoma%20patients%20in%20Canada